CLINICAL TRIAL: NCT05223829
Title: Utility of Brexanolone to Target Stress-induced Alcohol Use Among Men and Women With Posttraumatic Stress Disorder
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Sage Therapeutics (Industry)
Responsible Party: Principal Investigator, Mackenzie Peltier, Assistant Professor of Psychiatry, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000031354; U54AA027989 (NIH)
Record Dates: First submitted 2022-01-12; First posted 2022-02-04 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: PTSD; Alcohol Use Disorder
Keywords: alcohol; brexanolone; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism | interventions — brexanolone

STUDY DESIGN:
Intervention Model Description: This project is a Phase 1 (open-label, single arm, proof of concept) laboratory design. It will investigate the feasibility and safety of administering brexanolone to men and women and collect preliminary data to understand brexanolone's efficacy to reduce stress-induced drinking in individuals with PTSD/AUD.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Brexanaolone (Experimental): In this single-arm study, participants will be administered brexanolone as a continuous IV infusion over 20 hours (titrated up to 90mcg/kg/hour).
  Interventions: Drug: Brexanolone

INTERVENTIONS:
Drug: Brexanolone — Brexanolone will be administered as a continuous IV infusion over 20 hours under medical observation
  Other Names: Zulresso

SUMMARY:
For this protocol, the investigators plan to collect pilot data to: 1. establish the feasibility and safety of administering brexanolone to individuals with concurrent Posttraumatic Stress Disorder (PTSD) and Alcohol Use Disorder (AUD).

DETAILED DESCRIPTION:
This project is a Phase 1 (open-label, single arm, proof of concept) laboratory design. It will investigate the feasibility and safety of administering brexanolone to men and women with PTSD/AUD.

Eligibility screening consists of an intake session and a physical exam. Subjects meeting eligibility criteria will be administered brexanolone as a continuous IV infusion over 20 hours. Participants will be monitored during infusion by medical personnel. Forty-eight hours following drug administration, participants will then complete a laboratory session.

During the laboratory session, personalized imagery (stress) will precede a 2 hour alcohol self-administration period. Subjects will then complete a follow-up period, including assessments of alcohol use, PTSD symptoms, and side effects weekly for the next 30 days.

Primary outcome measures include treatment-emergent adverse events following administration of brexanolone for 30-days, as well as the percentage of milliliters consumed during ad-libitum drinking in the laboratory session. Additionally, at each visit the participants will complete a timeline follow-back assessment for a 30-day period (or the number of days in between intake, drug, and laboratory sessions) to explore a sustained reduction in in-vivo alcohol use.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 21-55 years old
4. Meet DSM-5 diagnostic criteria for AUD within the past 6 months, as well as the following drinking criteria:

   1. Men: drink greater than 14 drinks per week and exceed five drinks per day at least once per week within the past 30 days
   2. Women: drink greater than 7 drinks per week and exceed four drinks per day at least once per week within the past 30 days
5. Meet DSM-5 diagnostic criteria for PTSD in the past 6 months

Exclusion Criteria:

1. Actively seeking treatment for AUD
2. Likely to experience clinically significant alcohol withdrawal during the study procedures (e.g., history of alcohol-related perceptual distortions/hallucinations, seizures, or Clinical Institute Withdrawal Assessment Scale score > 8 at intake)
3. Current (i.e., past month) active suicidal ideation and/or homicidal ideation
4. Meets DSM-5 diagnostic criteria for schizophrenia, bipolar disorder, and/or other severe mental illnesses.
5. Meets criteria for current (past 6 months) substance use disorders (other than tobacco use disorder).
6. Tests positive for illicit substances during urine toxicology screens (except cannabis) at intake session
7. Is actively engaged in psychotherapy to treat PTSD
8. Any significant current medical conditions (neurological, cardiovascular [including hypertension or hypotension: sitting BP >160/100 or <90/60mmHg at baseline screening], endocrine, thyroid, renal, liver), seizures, delirium or hallucinations, or other unstable medical conditions including HIV
9. Past 30 day use of psychoactive drugs including anxiolytics and antidepressants.
10. Women who are pregnant or nursing, or fail to use one of the following methods of birth control unless she or her partner is surgically sterile or she is postmenopausal (hormone contraceptives [oral, implant, injection, patch, or ring], contraceptive sponge, double barrier [diaphragm or condom plus spermicide], or IUD)
11. Specific exclusions for the administration of brexanolone not already specified include: Individuals with end stage renal disease, treatment with any opioids or other CNS depressants, such as benzodiazepines.
12. Subjects likely to exhibit clinically significant alcohol withdrawal during the study. Specifically, we will exclude subjects who a) have a history of perceptual distortions, seizures, delirium, or hallucinations upon withdrawal or b) have a score of > 8 on the Clinical Institute Withdrawal Assessment scale at intake appointments.
13. Participation within the past 8 weeks in other studies that involve additive blood sampling and/or interventional measures that would be considered excessive in combination with the current application

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events | 30 days following administration of brexanolone
  Treatment-emergent adverse events will be assessed following administration of brexanolone.

CONTACTS AND LOCATIONS:
Overall Officials: MacKenzie R Peltier, PhD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No